CLINICAL TRIAL: NCT05778812
Title: A Study on Online Insomnia Treatment Programs
Brief Title: Online Insomnia Treatment Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Koko Home, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67436
Record Dates: First submitted 2023-03-10; First posted 2023-03-21 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Insomnia; Sleep; Sleep Disturbance; Sleep Disorder; Sleep Hygiene; Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias; Sleep Wake Disorders; Sleep Hygiene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full Sleep (Experimental): With Full Sleep, the app provides daily lessons about sleep and skills that can help with sleep. In the app, participants also record information about each night's sleep in their sleep log. Every seven nights, they also complete the Sleep Needs Questionnaire. At the beginning, middle, and end of the study, they additionally complete the Insomnia Severity Inventory in the app. At the end of every week, a sleep schedule and weekly summary are calculated via automated formulas. The app also contains access to messaging a coach. The intent of coach access is for participants to ask questions about their daily lessons and application of the skills and to feel supported and accountable.
  The REST (Radar Enabled Sensing Technology) device in the Full Sleep program uses radar to passively track sleep patterns and nighttime awakenings. It also offers white noise options and audio guidance for relaxation techniques and stimulus control.
  Interventions: Behavioral: Full Sleep
- Path to Better Sleep (Active Comparator): Path to Better Sleep is a self-management tool for insomnia. It is available as a web-based program at https://www.veterantraining.va.gov/apps/insomnia/index.html#dashboard. Path to Better Sleep is intended to be completed over six weeks, and includes weekly educational lessons about sleep which include videos, visual depictions, and interactive activities, in addition to sleep check-ins (e.g., knowledge checks, self reflections about sleep). It also includes sleep logging. Participants in this condition will be asked to share their sleep log weekly via email, as Stanford and Koko Labs do not receive access to the data.
  Interventions: Behavioral: Path to Better Sleep

INTERVENTIONS:
Behavioral: Full Sleep — Daily lessons about sleep and skills that can help with sleep. Participants also record information about each night's sleep in their sleep log. Every seven nights, they also complete the Sleep Needs Questionnaire. At the beginning, middle, and end of the study, they complete the Insomnia Severity Inventory in the app. At the end of every week, a sleep schedule and weekly summary are calculated via automated formulas. The app also contains access to messaging a coach, for participants to ask questions about their daily lessons and application of the skills and to feel supported and accountable.
  The REST device in the Full Sleep program uses radar to passively track sleep patterns and nighttime awakenings. It also offers white noise options and audio guidance for relaxation techniques and stimulus control.
  Arms: Full Sleep
Behavioral: Path to Better Sleep — Path to Better Sleep is a self-management tool for insomnia. It is available as a web-based program at https://www.veterantraining.va.gov/apps/insomnia/index.html#dashboard. Path to Better Sleep is intended to be completed over six weeks, and includes weekly educational lessons about sleep which include videos, visual depictions, and interactive activities, in addition to sleep check-ins (e.g., knowledge checks, self reflections about sleep). It also includes sleep logging. Participants in this condition will be asked to share their sleep log weekly via email, as Stanford and Koko Labs do not receive access to the data.
  Arms: Path to Better Sleep

SUMMARY:
The purpose of this study is to investigate improvements in sleep by comparing two 6-week digital programs, either online or app-based, that deliver Cognitive Behavioral Therapy for Insomnia (CBT-I), the "gold standard" treatment for insomnia, with or without a bedside device to help track sleep.

DETAILED DESCRIPTION:
Time needed from participant: 15 minutes per day to complete an app-based or online sleep diary and review information in an app-based or online CBT-I program.

To qualify, you must:

Be 18+ years old Have a diagnosis of insomnia or suspected insomnia Have access to the internet and an iphone, Android or other smart phone device

Coordinator Contact:

Cris Moreno (650) 721-7576 crismore@stanford.edu

ELIGIBILITY:
Inclusion Criteria:

* insomnia diagnosis or measure-confirmed moderate to severity insomnia (Insomnia Severity Index = 15-28)
* access to an iPhone with iOS 11+ or Samsung, Google, HTC, LG, OnePlus, or Motorola phone with Android 10+
* 18 years of age or older
* available 15 mins per day to participate

Exclusion Criteria:

* Restless Legs Syndrome
* narcolepsy
* sleep apnea
* sleep walking
* bipolar disorder
* seizures disorder
* substance abuse
* frailty/risk of falling
* severe memory problems
* shift work
* change in antidepressant medication within past 2 months
* serious mental/physical health problem
* other ongoing psychological treatment w
* sleeping with pets.

Participants should be aware that should they receive a device, its sound and light alerts could be disruptive to partners or others (e.g., children) that sleep in the same room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | Completion of program (6-8 weeks)
  A measure of insomnia symptoms

SECONDARY OUTCOMES:
Sleep efficiency | Completion of program (6-8 weeks)
  The proportion of time sleeping while in bed
Wakefulness after sleep onset | Completion of program (6-8 weeks)
  # minutes awake after falling asleep
Number of awakenings | Completion of program (6-8 weeks)
Sleep onset latency | Completion of program (6-8 weeks)
  Minutes to fall asleep
Total sleep time | Completion of program (6-8 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Sleep Medicine Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No